CLINICAL TRIAL: NCT06343350
Title: Prospective Pilot Study to Assess the Usability and Feasibility of OPTDR01 As an Automated Diabetic Retinopathy Screening Tool
Brief Title: OPTDR01 Feasibility for Automated Diabetic Retinopathy Detection
Status: Recruiting | Type: Observational
Sponsor: Optain Health (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTDR01P
Record Dates: First submitted 2024-03-25; First posted 2024-04-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy; Diabetes
Keywords: Artificial Intelligence; Diabetic Retinopathy; SaMD; Screening
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Retinal imaging: Participants will undergo retinal imaging with and without mydriatic agent to dilate the pupils.
  Interventions: Device: OPTDR01 software application

INTERVENTIONS:
Device: OPTDR01 software application — Retinal images will be sent to the OPTDR01 software application for mtmDR and vtDR detection

SUMMARY:
In the United States, only 62% of the 37 million people with diabetes receive annual screening exams for diabetic retinopathy. One of the goals of the US Department of Health and Human Services Healthy People 2030 campaign is to increase diabetic retinopathy screening rates to 70.3%. Research indicates that low screening rates are associated with a variety of factors, including income levels, race and lack of access to care. Furthermore, because diabetic retinopathy frequently presents asymptomatically, non-adherence to screening results in postponed disease detection and a higher probability of vision loss. Currently, it is estimated that 9 million adults in the US are affected by diabetic retinopathy, and 1.8 million suffer from vision-threatening diabetic retinopathy. Importantly, the rates of vtDR vary greatly by race, with Hispanic individuals at 7.14% and Black individuals at 8.66%, compared to 3.55% in White individuals. Despite these alarming figures, the disease can be managed and vision loss can often be averted with early disease detection, thus highlighting the importance of increasing screening rates.

A clear need exists for a diabetic retinopathy screening tool that can be deployed in primary care settings, addressing the shortage of specialist care and making screening more accessible to underserved populations. OPTDR01 will directly address these issues by providing accessible, high quality screening for diabetic retinopathy. OPTDR01 will automatically detect more than mild diabetic retinopathy (mtmDR) and vision-threatening diabetic retinopathy (vtDR) in diabetic adults who have not previously been diagnosed with mtmDR or vtDR.

DETAILED DESCRIPTION:
This study will be conducted to assess the feasibility of the OPTDR01 in detecting mtmDR and vtDR in frontline care settings in adults with a diagnosis of diabetes but no prior diagnosis of diabetic retinopathy. The study will inform the design of a large pivotal study in terms of expected disease prevalence, participant recruitment rate, data collection tools and study workflow.

Eligible participants will undergo the following:

* retinal imaging sessions of each eye with a fundus camera for OPTDR01 evaluation
* dilation with mydriatic agent
* fundus photography, macular optical coherence tomography (OCT) and red reflex exam of each eye for comparison.

A subset of participants will be invited to participate in a precision sub-study, during which multiple operators will image participant eyes with multiple cameras.

ELIGIBILITY:
Inclusion Criteria:

1. Having met the criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA):
2. Age 22 or older
3. Understand the study and volunteer to sign the informed consent

Exclusion Criteria:

1. Unable to understand the study
2. Unwilling to sign informed consent
3. Indicate persistent vision loss, blurred vision, or floaters
4. Previous diagnosis of macular edema, diabetic retinopathy (any level) proliferative retinopathy, radiation retinopathy, or retinal vein occlusion
5. History of laser treatment of the retina or injections into either eye, or any history of retinal surgery
6. Currently participating in another investigational eye study or actively receiving investigational product for diabetic retinopathy or diabetic macular edema
7. A condition that, in the opinion of the investigator, would preclude participation in the study
8. Contraindicated for imaging by fundus imaging systems used in the study because of hypersensitivity to light, recently underwent photodynamic therapy, or was taking medication that causes photosensitivity
9. Known pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Type I or Type II diabetes that are eligible for Diabetic Retinopathy screening
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate of eligible participants at clinical site | Assessed weekly until study end
  Number of eligible participants that are enrolled on a weekly basis at a clinical site

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Gastro SB, Chula Vista, California
  - Triwest Research Associates, San Diego, California
  - Precision Research Institute, San Diego, California
  - Gulf Coast Clinical Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No